CLINICAL TRIAL: NCT02107768
Title: Effects of Twice-Weekly Intense Aerobic Exercise in Early Subacute Stroke: A Randomized Controlled Trial.
Brief Title: Aerobic Exercise in Early Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klas Sandberg (Other)
Responsible Party: Sponsor-Investigator, Klas Sandberg, MSc,RPT, Ostergotland County Council, Sweden
Organization: Ostergotland County Council, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/396-31
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Stroke
Keywords: Stroke; Exercise; Randomized trial; Quality of Life
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise recommendation (Experimental): Patients randomized to the control group receive general advice for physical training and activity but no specific training or other rehabilitation efforts
  Interventions: Other: Aerobic exercise
- Aerobic exercise (Experimental): The intervention group will conduct a 12 week training period with two training sessions of 60 minutes per week at a local hospital. The start shall be made within 6 weeks after stroke . The training shall be conducted in a group with a maximum of 10 participants and start running as new participants in the intervention group will be added. The intensity during the exercise program should be individualized and based on the initial tests . Patients should be advised to reach a degree of exertion 13-15/20, Rate of Perceived Exertion (Borg 's RPE scale)
  Two fitness goals was to be achieved during the training session:
  1. An individual training level corresponded to 50% or more of maximal oxygen uptake for at least 40 min ( Borg 9-11/20 ) . Which corresponds to 70 % of maximum heart rate.
  2:nd 80% or more of the estimated maximum oxygen uptake during two periods of 8 minutes( Borg 13-15/20 ) .Which corresponds to 85% of maximum heart rate.
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — Other: Aerobic exercise The intervention group will conduct a 12 week training period with two training sessions of 60 minutes per week at a local hospital. The start shall be made within 6 weeks after stroke . The training shall be conducted in a group with a maximum of 10 participants and start running as new participants in the intervention group will be added.The intensity during the exercise program should be individualized and based on the initial tests . Patients should be advised to reach a degree of exertion 13-15/20,Rate of Perceived Exertion (Borg 's RPE scale) .
  Two fitness goals was to be achieved during the training session
  1. An individual training level corresponded to 50% or more of maximal oxygen uptake for at least 40 min ( Borg 9-11/20 ) . Which corresponds to 70 % of maximum heart rate.
  2:nd 80% or more of the estimated maximum oxygen uptake during two periods of 8 minutes( Borg 13-15/20 ) . Which corresponds to 85 % of maximum heart rate.

SUMMARY:
The purpose of this study was to investigate the effects of early intensive aerobic exercise regarding aerobic capacity, gait and balance, Health Related Quality of Life and participation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand Swedish language.
* Ability to walk 5 meters with or without the support of any means or person.
* Be able to get up on a cycle ergometer and cycle in their own chosen pace.
* Approval of medically responsible physician to conduct physical training in groups.

Exclusion Criteria:

* Medical or neurological diseases that may affect the exercise execution.
* Patients for whom transportation to and from hospital can not be arranged during intervention period

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity | Baseline,3month
  cardiorespiratory stress test (Watt)

SECONDARY OUTCOMES:
Balance | Baseline,3month
  Time Up and Go(TUG) ,Single Leg Stance(SLS)
Walking capacity | Baseline,3month
  Six minute walk test (6MWT ), 10 meters Walking test

OTHER OUTCOMES:
EQ5-D | Baseline,3month,6month
  Quality of life
Stroke Impact Scale | Baseline,3month,6month
  Recovery after stroke, participation

CONTACTS AND LOCATIONS:
Overall Officials: Klas Sandberg, Msc,RPT, Principal Investigator — Rehab East, Local Health Care Östergötland County Council; Marie Kleist, Bsc,RPT, Principal Investigator — Rehab East, Local Health Care Östergötland County Council; Lars Falk, PhD,MD, Principal Investigator — Research and Development Unit, Local Health Care Östergötland County Council, Dept of Dermatology and Venereology, Linköping University Hospital,; Paul Enthoven, PhD,RPT, Principal Investigator — Research and Development Unit, Local Health Care Östergötland County Council,Dept of Medical and Health Sciences, Linköping University

REFERENCES:
- [Derived] Wijkman MO, Sandberg K, Kleist M, Falk L, Enthoven P. The exaggerated blood pressure response to exercise in the sub-acute phase after stroke is not affected by aerobic exercise. J Clin Hypertens (Greenwich). 2018 Jan;20(1):56-64. doi: 10.1111/jch.13157. Epub 2018 Jan 16. PMID 29338111
- [Derived] Sandberg K, Kleist M, Falk L, Enthoven P. Effects of Twice-Weekly Intense Aerobic Exercise in Early Subacute Stroke: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 Aug;97(8):1244-53. doi: 10.1016/j.apmr.2016.01.030. Epub 2016 Feb 20. PMID 26903147